CLINICAL TRIAL: NCT07228078
Title: An Open-Label Extension (OLE) Study to Evaluate the Long-Term Safety, Tolerability and Exploratory Efficacy of SNK01 in Participants With Alzheimer's Disease (Study SNK01-AD02)
Brief Title: Open-Label Extension Protocol to SNK01-AD01 Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NKGen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNK01-AD02
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
Keywords: Moderate Alzheimer's Disease; AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label (Experimental): SNK01
  Interventions: Biological: SNK01

INTERVENTIONS:
Biological: SNK01 — SNK01 is a novel cell-based, patient specific ex vivo expanded autologous natural killer (NK) cell, immunotherapeutic drug

SUMMARY:
Open-Label Extension Protocol to SNK01-AD01 Study

DETAILED DESCRIPTION:
Open-label extension study to assess long-term safety and tolerability of SNK01 administered as an intravenous (IV) infusion every 3 weeks in participants with Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

Participants will be considered eligible for participation in the study if all the following criteria are satisfied:

* The participant or their legally authorized representative must be willing and able to give their informed consent in writing and comply with the requirements of this study protocol. Informed consent for participants or their legally authorized representative and caregivers will be obtained before any trial-related activity. (Trial-related activities are any procedure that would not be performed during normal treatment of the subject).
* Participants must have a reliable study partner/caregiver (per investigator judgement for instance a family member, partner etc., guardian (must be always the same person)) who is in close contact with the patient, available on call and who is able to contribute to the assessment of the ratings of the functional endpoints at specific study visits. This person will be able to communicate in the language in which the participant is being assessed and should also serve as a backup contact for the study site.
* Participants previously completed participation in study SNK01-AD01.

Exclusion Criteria:

Participants who fulfill any of the following criteria will not be recruited into the study:

• Any participant whose safety the investigator considers to be at risk from this trial's intervention.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1 Year
  Evaluate the safety and tolerability of SNK01 assessed by labs, PE and AEs

SECONDARY OUTCOMES:
Preliminary efficacy in cognitive assessment scores of CDR-SB | 1 Year
  Measure changes in cognitive assessment of CDR-SB from baseline
Preliminary efficacy in cognitive assessment scores of MMSE | 1 Year
  Measure changes in cognitive assessment of MMSE from baseline
Preliminary efficacy in cognitive assessment scores of NPI | 1 Year
  Measure changes in cognitive assessment of NPI from baseline
Preliminary efficacy in cognitive assessment scores of ADCS-ADL-Severe | 1 Year
  Measure changes in cognitive assessment of ADCS-ADL-Severe from baseline
Preliminary efficacy in cognitive assessment scores of ADAS-Cog | 1 Year
  Measure changes in cognitive assessment of ADAS-Cog from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioral Research Specialists, LLC, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No